CLINICAL TRIAL: NCT00038363
Title: Comparison of Subacute and Hospital Based Rehabilitation Care
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: O2571R
Record Dates: First submitted 2002-05-30; First posted 2002-05-31 (Estimated); Last update posted 2009-01-21 (Estimated); Status verified 2002-05

CONDITIONS: Aging
Keywords: Frail; Disable; Disabled Persons; Physically disabled; Elderly; Rehabilitation; Subacute care
MeSH Terms: interventions — Rehabilitation; Subacute Care

INTERVENTIONS:
Procedure: Rehabilitation
Procedure: Subacute care

SUMMARY:
The proposed study objective is to compare hospital-based rehabilitative care with transitional subacute rehabilitation for adults recently diagnosed with a disabling disorder. Clinical outcomes, cost and utilization of services will be compared in order to test the hypotheses that medically-stable patients receiving rehabilitation from subacute care facilities will: 1) function as well physically, 2) report less family dysfunction, 3) have better psychological adjustment and well-being than controls who receive only hospital-based inpatient care, and 4) receive services at lower cost. We intend to assess the impact of hospital-based versus subacute care on clinical and cost outcomes at admission, discharge [3 months post-admission] and at 12 months. The first set of analyses will determine predictors of physical function, family function, psychological adjustment and well-being over a 1 year period.

DETAILED DESCRIPTION:
Although subacute transitional care is thought to reduce costs by as much as 60 percent of hospital-based care costs (DHHS, 1995), systematic prospective studies of utilization and cost of services have not been done. An important factor to be considered, particularly in elderly patients, is the cost associated with readmission. Some studies have suggested that cost savings and reduced readmissions are associated with the increased availability of post-discharge services (Ludke, MacDowell, Booth et. al., 1990; Weinberger, Smith, Katz et al., 1988). If such cost savings exist, then transitional subacute care may be an important community-based resource for patients returning to independent living. In addition to demonstrating the clinical efficacy of subacute transitional care, the proposed study will also assess long-term outcomes, taking into account patient resource utilization and the incidence of readmission.

The current study will determine if subacute transitional care can improve outcomes that are important to the broad goals of long term independent living and enhanced quality of life. Variables assessed will focus on physical and family function, adjustment, resource utilization, skilled care placements, and survival. When compared to hospital-based rehabilitation, subacute rehabilitation is expected to demonstrate improvements in physical abilities, family function, adjustment, well being, and survival.

b. Hypothesis. The primary hypothesis is that clinical outcomes will be significantly better for subacute care patients at 3 and 12 months than hospital-based control patients. Costs and resource utilization are hypothesized to be significantly less.

c. Objectives and projected timeline. The objective of this study is to conduct a randomized clinical trial to examine the effects of subacute transitional care compared with hospital-based rehabilitative care for disabled patients. Specific objectives will be to: 1] evaluate the type, magnitude and duration of rehabilitative care provided, 2] determine differences in cost of care provided to the two groups, 3] compare clinical outcomes of the two treatments by assessing the magnitude of change, and 4] compare long-term outcomes at 12 months.

Secondary objectives will be to describe diagnostic or demographic subgroups who may benefit to a greater or lesser extent than others.

Patients will be recruited into the study and followed for 1 year, with measurements occurring at hospital admission, at 3 months, and at 12 months. The time to completion of the study is projected to be 3 years. Recruitment of subjects will begin during the second quarter of the project and will continue for 1.5 years. Follow-up measures will continue for an additional year.

ELIGIBILITY:
Disabling disorders

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 260 (Estimated)
Dates: Start 2001-04; Study Completion 2004-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Wolff, Ph.D. Special Assistant to the Director — Program Analysis and Review Section (PARS), VA Rehabilitation Research & Development Service; Vicki Mongiardo, Program Analyst — Program Analysis and Review Section (PARS), VA Rehabilitation Research and Development Service
Locations (1):
- VA Medical Center, Seattle, Washington, United States